CLINICAL TRIAL: NCT01495078
Title: Telemonitoring and Teleintervention of Heart Failure and Decrease of Non-fatal Events.
Acronym: ICOR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Parc de Salut Mar (Other)
Responsible Party: Principal Investigator, Josep Comín, Josep Comin-Colet, Parc de Salut Mar
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Proyecto ICOR
Record Dates: First submitted 2011-09-08; First posted 2011-12-19 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2016-02

CONDITIONS: Heart Failure
Keywords: telemonitoring; heart failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Telemonitoring (Experimental): Patients with follow-up telemonitoring
  Interventions: Procedure: Telemonitoring
- Non - telemonitoring (No Intervention): Patients with usual face follow-up

INTERVENTIONS:
Procedure: Telemonitoring — Is a computer system designed jointly by engineers and clinical personal of Parc Salut Mar) to be able daily automated selfreported symptom and weight, blood pressure and heart rate monitoring . The system allow weekly follow up throught videoconferences.
  Information from the telemonitoring system is automatically downloaded to a secure Internet site for review by clinicians and nurses.
  Arms: Telemonitoring

SUMMARY:
The primary objective of the study is to determine the effect of automated daily selfreported symptom and weight, blood pressure and heart rate monitoring and clinical follow-up videoconference comigrate with clinical follow-up face in specialized hospital unit in reducing heart failure non-fatal events.

DETAILED DESCRIPTION:
The insuﬁcie 'ncia Cardı´aca Optimitzacio ´ Remota (iCOR; Heart Failure Remote Optimization) trial was a singlecentre, randomized, open-label study designed to evaluate the eﬃcacy of the addition of telemedicine (telemonitorization and teleintervention using videoconference) to an existing specialized, multidisciplinary, nurse-based, hospitalprimary care integrated HF programme for high-risk patients with CHF. The organizational characteristics of the programme and the impact in health outcomes resulting from its implementation have been previously published.2 In this study we aimed to compare the strategy of providing nurse-based structured follow-up to high-risk CHF patients through planned contacts between health care providers and patients and/or caregivers in the basis of face-to-face on-site encounters (usual care in our HF programme) or provide the planned care using telemedicine with the combination of remote daily monitoring of signs and symptoms of HF (telemonitoring) and delivery of structured nursebased follow-up health care using videoconference (teleintervention). The main hypothesis of this study was that adding telemedicine to an existing HF programme would be associated with a reduction in the number of non-fatal HF events in high-risk patients with CHF. As a secondary hypothesis we assumed that adding telemedicine would translate into a reduction in health care resource utilization and subsequently in health care costs.

ELIGIBILITY:
Inclusion Criteria:

* Patients discharged from a heart failure hospitalization within 30 days of enrollment into the study.

Exclusion Criteria:

* Less than 18 years
* Long-term nursing home residence, irreversible medical conditions, Folstein Mini-mental State Exam score less than 20.
* No access to 3G line, currently scheduled for cardiac transplant, left ventricular assist device or valvular surgery,coronary intervention within 90 days of randomisation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2010-12; Primary Completion 2013-06 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Non fatal events | Six months after inclusion of the patient.
  Non fatal events are defined as an event of descompensation requiring either parenteral treatment as outpatients in a day hospital an in the emergency department or by income.

SECONDARY OUTCOMES:
Morbid mortality | From telemonitoring (baseline) until six months later
Hospital readmission | From telemonitoring (baseline) until six months later

CONTACTS AND LOCATIONS:
Overall Officials: JOSEP COMIN COLET, MD, Principal Investigator — HOSPITAL DEL MAR MEDICAL RESEARCH INSTITUTE
Locations (1):
- Parc de Salut Mar, Barcelona, Spain, Spain

IPD SHARING:
Plan to Share IPD: No